CLINICAL TRIAL: NCT06326190
Title: 177Lu-DOTATATE for Recurrent Meningioma: a Randomized Phase II Study
Brief Title: 177Lu-DOTATATE for Recurrent Meningioma
Acronym: LUMEN-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-2334-BTG
Record Dates: First submitted 2024-03-14; First posted 2024-03-22 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Meningioma
Keywords: 177Lu-DOTATATE; Meningioma; Recurrent Meningioma; Phase II
MeSH Terms: conditions — Meningioma | interventions — Hydroxyurea; Bevacizumab; Sunitinib; Octreotide; Everolimus; Observation; lutetium Lu 177 dotatate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group: local standard of care (LOC) (Active Comparator): According to local standard practice, treatment in the control arm is left to the investigator's discretion.
  * Hydroxyurea
  * Bevacizumab
  * Sunitinib
  * Octreotide (Sandostatin LAR)
  * Everolimus
  * No treatment (observation with regular follow-up and best supportive care)
  Interventions: Drug: Local standard of Care
- Experimental group: 177Lu-DOTATATE (Experimental): Patients will receive 177Lu-DOTATATE with a total dose of 7.4 GBq/cycle every four (4) weeks for four (4) cycles as an IV infusion
  Interventions: Drug: 177Lu-DOTATATE

INTERVENTIONS:
Drug: Local standard of Care — According to local standard practice, treatment or no treatment in the control arm is left to the investigator's discretion.
  Other Names: Hydroxycarbamide; Bevacizumab; Sunitinib; Octreotide (Sandostatin LAR); Everolimus; No active treatment (observation with regular follow-up and best supportive care)
  Arms: Control group: local standard of care (LOC)
Drug: 177Lu-DOTATATE — Intravenous injection of 177Lu-DOTATATE
  Other Names: ¹⁷⁷Lu-DOTA0-TATE; Lutathera®; Lu oxodotreotide
  Arms: Experimental group: 177Lu-DOTATATE

SUMMARY:
Novel treatments are urgently needed for meningiomas progressing after local therapies (surgery, radiotherapy). So far, no effective systemic therapies are known in this situation. The LUMEN-1 trial will investigate in a prospective randomized trial the efficacy of the precision medicine "theranostic" concept of combining diagnostic patient selection using PET-based molecular imaging and target-specific therapeutic intervention using a systemically administered radioligand.

The rationale for the LUMEN-1 trial is based on the following: (a) high somatostatin receptor (SSTR) expression in meningiomas, (b) wide-spread availability of clinically established SSTR-PET imaging, (c) proven efficacy of SSTR-targeting radioligand therapy using [177Lu]Lu-DOTATATE in another tumor type (neuroendocrine tumors), and (d) promising experiences with [177Lu]Lu-DOTATATE therapy in compassionate use applications and retrospective case series and interim results from one ongoing uncontrolled prospective trial in meningiomas. LUMEN-1 is the first randomized clinical trial to investigate [177Lu]Lu-DOTATATE therapy in refractory meningioma and may open new avenues for treatment and research in this area.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥ 18 years of age
* Histologically confirmed diagnosis of meningioma (all grades, 1-3 per WHO CNS5, are eligible)
* WHO performance status 0-2
* Measurable disease (at least 10 x10 mm contrast enhancing lesion) on cranial MRI no more than two weeks prior to randomization
* Radiologically documented progression of any existing tumour (growth > 25% in the last two years) or appearance of new lesions (including intra- and extracranial manifestations)
* Somatostatin receptor (SSTR)-positive confirmed by PET imaging with scan performed within four weeks before randomization (baseline SSTR-PET is considered as positive when meningioma uptake intensity exceeds a SUVmax of 2.3).
* At least one prior surgery and one line of external beam radiotherapy for meningioma
* Adequate liver, renal and haematological function within four weeks prior to randomization (1) Neutrophils ≥ 1.5 x 109/L, hemoglobin ≥ 9 g/dL or hemoglobin ≥ 5.6 mmol/L, platelets ≥ 100 x 109/L, (2) Total Bilirubin ≤ 1 x ULN, SGPT/ALT and SGOT/AST ≤ 2.5 x ULN, (3) Albumin ≥ 30 g/L, (4) Serum creatinine ≤ 1.5 x ULN, (5) Creatinine clearance > 40 ml/min as calculated by CKD-EPI 2021
* Participants must have the following electrolyte values within normal limits or corrected to be within normal limits with supplements prior to first dose of study medication: (1) Potassium (potassium level of up to 6.0 mmol/L is acceptable at study entry if associated with creatinine clearance within normal limits calculated using CKD-EPI formula). Mild decrease below lower limit of normal (LLN) is acceptable at study entry if considered not clinically significant by investigator, (2) Magnesium, with the exception of magnesium level > ULN - 3.0 mg/dL (1.23 mmol/L) associated with creatinine clearance within normal limits calculated using CKD-EPI formula. Mild decrease below LLN is acceptable at study entry if considered not clinically significant by Investigator, (3) Total calcium (corrected for serum albumin) level of up to 12.5 mg/dL (3.1 mmol/L) is acceptable at study entry if associated with creatinine clearance within normal limits calculated using CKD-EPI formula. Mild decrease below LLN is acceptable at study entry if considered not clinically significant by Investigator.
* Patients who are receiving corticosteroid treatment with dexamethasone, must be treated with a dose of ≤4 mg/day (or other corticosteroids equivalent dose) for a minimum of 7 days initiation of study treatment.
* Women of childbearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 72 hours prior to randomization. A positive urine pregnancy test result must immediately be confirmed using a serum test. A pregnancy test is to be reported within 7 days prior to the first dose of the study treatment. Note: women of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e., females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrhoeic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antioestrogens, low body weight, ovarian suppression, or other reasons.
* Patients of childbearing / reproductive potential should use adequate birth control measures during the study treatment period and for at least 6 months after the last dose of treatment. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. Such methods include: (1) Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), (2) Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), (3) Intrauterine device (IUD), (4) Intrauterine hormone-releasing system (IUS), (5) Bilateral tubal occlusion, (6) Vasectomized partner, (7) Sexual abstinence (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient)
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 7 months after the last study treatment.
* Before patient 's enrolment, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Local therapy (surgery and / or radiotherapy) indicated per local investigator. Note: in case of patients with multiple meningioma lesions, in whom resection and / or radiotherapy of individual lesions is indicated, patients may be included after local therapy (with a 4-week gap between surgery / end of radiotherapy and start of treatment), if at least one remaining lesion fulfils the inclusion criteria.
* Any combined or any prior systemic treatment regardless the timing.
* Life expectancy is less than nine weeks.
* History of any other invasive malignancy within the last five years (except adequately treated non-melanoma skin cancer, clinically localized and very low-risk prostate cancer, and adequately treated cervical intraepithelial neoplasia)
* Suspected pregnancy or when pregnancy has not been excluded
* Contraindication to MRI, CT or PET
* Unstable cardiac conditions (congestive heart failure, angina pectoris, myocardial infarction within one year before randomization, uncontrolled hypertension, clinically significant arrhythmias)
* Psychological, familial, sociological, or geographical conditions potentially hamper compliance with the study protocol and follow-up schedule.
* Known hypersensitivity to the active substance or to any excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-04-14 (Estimated); Study Completion 2028-12-22 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | From the date of randomization till the date of disease progression or death (time till death is up to 2 years after patient enrolment in the study)
  To examine whether [177Lu]Lu-DOTATATE demonstrates sufficient antitumor activity in patients with recurrent meningioma to justify further investigation. Progression-free survival computed based on MRI-based RANO meningioma response criteria as assessed by the local investigator.

SECONDARY OUTCOMES:
Overall Survival (OS) | From the date of randomization till the date of death (time till death is up to 2 years after patient enrolment in the study)
  Overall survival (OS), OS probability at 6 (OS6) and 12 months (OS12), median OS (mOS)
Radiological response rate | From the date of randomization till the date of disease progression or death (time till death is up to 2 years after patient enrolment in the study)
  Best overall response (BOR, defined as CR, MR or PR during study treatment) rate. Complete response (CR) rate is computed by MRI based RANO meningioma response criteria as assessed by the local investigator.
Radiological response rate | From the date of randomization till the date of disease progression or death (time till death is up to 2 years after patient enrolment in the study)
  Median best overall response (BOR, defined as CR, MR or PR during study treatment) duration. Median complete response (CR) duration is computed by MRI based RANO meningioma response criteria as assessed by the local investigator.
The magnitude of change in Health-related quality of life (HRQoL) | From the date of randomization regardless of progression status up to 2 years after patient enrolment in the study.
  The magnitude of change in HRQoL in terms of global health status from EORTC QLQ-C30 during treatment.
The magnitude of change in Health-related quality of life (HRQoL) | From the date of randomization regardless of progression status up to 2 years after patient enrolment in the study.
  The magnitude of change in HRQoL in terms of physical functioning from EORTC QLQ-C30 during treatment.
The magnitude of change in Health-related quality of life (HRQoL) | From the date of randomization regardless of progression status up to 2 years after patient enrolment in the study.
  The magnitude of change in HRQoL in terms of motor disfunction from EORTC QLQ-BN20 during treatment.
Neurological function (NANO scale) | From the date of randomization regardless of progression status up to 2 years after patient enrolment in the study.
  Change of neurological function (NANO scale) from baseline during study treatment.
Toxicity According to CTCAE Version 5.0 | From the date of randomization regardless of progression status up to 2 years after patient enrolment in the study.
  This study will use the International Common Terminology Criteria for Adverse Events (CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Nathalie Albert, Principal Investigator — EORTC Study Coordinator
Locations (12):
- Austria (2):
  - A.O Landeskrankenhaus - Innsbruck Universitaetsklinik, Innsbruck
  - Universitaetskliniken der Uni Wien - Universitaetsklinikum Wien - AKH unikliniken, Vienna
- France (4):
  - Centre Leon Berard, Lyon
  - Centre Eugene Marquis, Rennes
  - CHRU de Nancy - Hopitaux De Brabois, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif
- Norway (2):
  - Oslo University Hospital - Radiumhospitalet, Oslo
  - St Olavs University Hospital - St. Olavs Hospital, Trondheim University Hospital, Trondheim
- Spain (2):
  - Vall D Hebron - Hospital Universitari Vall d'Hebron -Vall d'Hebron Institut Oncologia, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
- Switzerland (2):
  - Oncology Institute of Southern Switzerland (IOSI) - Ospedale San Giovanni, Bellinzona
  - UniversitaetsSpital Zurich - Neurology Clinic, Zurich